CLINICAL TRIAL: NCT05044689
Title: Case Control Study to Identify Modifiable Risk Factors for Colorectal and Breast Cancer in Nigeria
Status: Recruiting | Type: Observational
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Lagos State University (Other); University of Ilorin Teaching Hospital (Other); Federal Medical Centre, Owo (Industry); University of Maiduguri Teaching Hospital (Unknown); National Hospital, Abuja (Other Government)
Responsible Party: Principal Investigator, Olusegun Alatise, MB.ChB (Ife), M.Sc, FWACS, FMCS, FACS, Obafemi Awolowo University Teaching Hospital
Other Study IDs: ERC/2018/06/01
Record Dates: First submitted 2021-09-09; First posted 2021-09-16 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Breast Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Colorectal Cancer (Cases): Based on the existing ARGO (African Colorectal Cancer Group) platform where a current colorectal cancer study is going on, 400 patients with a prior diagnosis and a new diagnosis will be recruited into this study.
  Interventions: Behavioral: Questionnaire; Device: Bioimpedance/Body Composition Unit
- Controls: We will select our 400 controls from two groups of participants who are free of cancer and gastrointestinal diseases. First, we will leverage community mobilization groups to identify and recruit a target group of 200 community-based population controls. Second, we will identify and recruit the remaining 200 controls from those seeking care in the Outpatient Health Center at OAU, which sees ~50-60 patients per day as part of routine care.
  Interventions: Behavioral: Questionnaire; Device: Bioimpedance/Body Composition Unit

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire containing questions regarding diet, physical activity, past medical history and life style practices.
Device: Bioimpedance/Body Composition Unit — Patients will provide information on body composition through the use of a bioimpedance machine which measures the body mass index, fat and total body water.

SUMMARY:
This project is a case-control study which seeks to identify modifiable risk factors for breast and colorectal cancer in Nigeria. Both cases and controls will be required to complete a risk factor questionnaire which contains information about their diet, physical activity, past medical history and life style factors. They will also be required to provide information on their body composition through the use of a bioimpedance machine which measures the body mass index, fat and total body water percentage.

Based on the existing ARGO platform where a current colorectal cancer study is going on, approximately 400 patients with a prior diagnosis or a new diagnosis will be recruited into this study. Comparatively, we will select our 400 controls from two groups of participants who are free of cancer and gastrointestinal diseases.

ELIGIBILITY:
Case Group - Patients must have histologically confirmed diagnosis of colorectal or breast cancer.

Control Group - Patients must not have a diagnosis of cancer.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Based on the existing African Research Group for Oncology platform where a current colorectal study is going on, 400 patients with a prior diagnosis and a new diagnosis of colorectal cancer or breast cancer will be recruited into this study.
  A combined total of 400 controls will be recruited from community mobilization groups and the Outpatient Health Center at OAU who are free of cancer and gastrointestinal diseases.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Development and Validation of Questionnaire For Assessing Modifiable Risk Factors for Cancer in Sub-Saharan Africa | 2 years
Determination of Novel Modifiable Cancer Risk Factors in a Nigerian Population | 2 years
  We will determine the presence of established, plausible, and novel cancer risk factors in cases (n=400) and controls (n=400) in Nigeria

CONTACTS AND LOCATIONS:
Locations (1):
- Obafemi Awolowo University Teaching Hospitals, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No